CLINICAL TRIAL: NCT02509416
Title: Rapid Assessment of Trainee Endoscopy Skills (RATES) Study Two: A Prospective Multicenter Study Evaluating Competence in Endoscopic Ultrasound and Endoscopic Retrograde Cholangiopancreatogram Among Advanced Endoscopy Trainees
Brief Title: Rapid Assessment of Trainee Endoscopy Skills (RATES) Study Two
Acronym: RATES 2
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: Columbia University (Other); Beth Israel Deaconess Medical Center (Other); Carolinas Medical Center (Other); The Cleveland Clinic (Other); Duke University (Other); Emory University (Other); Geisinger Clinic (Other); St. Luke's Medical Center (Other); Johns Hopkins University (Other); Northwestern University Feinberg School of Medicine (Other); Stanford University (Other); Stony Brook University (Other); University Hospitals Cleveland Medical Center (Other); University of Alberta (Other); University of California, Los Angeles (Other); University of Florida (Other); University of Massachusetts, Worcester (Other); University of Michigan (Other); University of Pennsylvania (Other); The University of Texas Health Science Center at San Antonio (Other); University of Texas (Other); University of Virginia (Other); Weill Medical College of Cornell University (Other); Brigham and Women's Hospital (Other); Dartmouth-Hitchcock Medical Center (Other); Virginia Mason Hospital/Medical Center (Other); Henry Ford Hospital (Other); Icahn School of Medicine at Mount Sinai (Other); Mayo Clinic (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); University of California, Davis (Other); Indiana University (Other); University of Kansas (Other); University of Wisconsin, Madison (Other); Vanderbilt University Medical Center (Other); Washington University School of Medicine (Other); University of North Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: 14-0604-2
Record Dates: First submitted 2015-07-01; First posted 2015-07-28 (Estimated); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Competency Based Education
Keywords: endoscopic ultrasound; endoscopic retrograde cholangiopancreatography; competency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The establishment of a number of training programs in therapeutic endoscopy, standardization of the performance of endoscopic ultrasound (EUS) and endoscopy retrograde cholangiopancreatography (ERCP) and definition of competence is of paramount importance. The length of training and minimum number of procedures, requisite theoretical learning and methodology to define competence in EUS and ERCP are not well defined. The investigators research has demonstrated that individuals in training acquire skills at different rates and the number of procedures completed alone is a suboptimal marker for competency in a given procedure. Hence, emphasis needs to be shifted away from the number of procedures performed to performance metrics with well-defined and validated thresholds of performance. Multicenter prospective data are needed to help guide development of competency based medical education that define learning curves in EUS and ERCP and set evidence-based benchmarks required to achieve competence using a validated competency assessment tool.

Hypothesis: The central hypothesis is that a validated EUS and ERCP competency assessment tool will allow for reliable and generalizable standardized learning curves, competency benchmarks and creation of a centralized national database that compares a trainee's performance amongst peers.

DETAILED DESCRIPTION:
Competency-based medical education and milestones: Given the increasing emphasis on quality metrics and competency in health care, the Accreditation Council for Graduate Medical Education (ACGME) recently announced plans to replace their current reporting system in 2014 with the Next Accreditation System (NAS). This reporting system focused on: 1) ensuring that milestones are reached at various points in training, 2) ensuring that competence is achieved by all trainees, and 3) making certain that these assessments are documented by their programs.

Learning curves and competence in EUS: EUS is a vital tool in the diagnosis and staging of gastrointestinal and certain non-gastrointestinal malignancies and diseases. EUS is operator dependent and training in EUS requires the development of technical and cognitive skills beyond that required for standard endoscopic procedures. It is intuitive that the quality of EUS in provision of patient care is directly proportional to the training, skill and experience of the endosonographer. Unfortunately, the intensity and length of training and minimum number of procedures required, requisite curriculum and extent of theoretical learning, and methodology to define competence are not well defined. There are limited data on learning curves in EUS imaging.Based on expert opinion, the American Society of Gastrointestinal Endoscopy (ASGE) recommends a minimum of 150 total supervised procedures, 75 of which have a pancreatobiliary indication and 50 cases of fine needle aspiration (FNA) (25 of which are pancreatic FNA) before competency can be determined.

Similar guidelines were recently proposed by the British Society of Gastroenterology (BSG)13 and the European Society of Gastrointestinal Endoscopy. However, these guidelines have not been validated. This does not account for the different rates at which people learn and in fact, many experts believe that the majority of trainees will require double the number of proposed procedures to achieve competency in EUS.

Learning curves and competence in ERCP: ERCP is an effective modality in the evaluation and management of pancreatobiliary diseases. This procedure can be technically demanding and associated with a wide range of adverse events. Technically failed ERCP may result in complications, need for additional procedures and their associated costs. Similar to EUS, ERCP is operator dependent and requires acquisition of certain technical and cognitive skills. There are limited data on learning curves and competence in ERCP, a cannulation rate of >80% (with some suggesting >90%) has been considered a surrogate for trainee competency. The ASGE recommends a minimum of 180 total procedures, the majority of which are therapeutic before competency can be achieved. However, this threshold is based predominantly on biliary cannulation success rate and does not take into account procedure complexity and the different rates at which people learn. It is also important to note that none of the previous studies have evaluated learning curves and competency in other quality indicators such as successful stone extraction, traversing and dilating a stricture, stent placement to name a few.

Competency assessment tools: Previous competency assessment tools have focused primarily on a limited number of motor skills involved in EUS and ERCP with no procedure-related cognitive skill assessment. The investigators have designed a prospective comprehensive competency assessment tool using validated benchmarks to define competency thresholds. The EUS and ERCP Skills Assessment Tool (TEESAT) can be used in a continuous fashion throughout the duration of training to grade technical and cognitive skills in EUS and ERCP in a balanced manner.

Significance, Innovation and Impact on Training and Education with the launch of the ACGME's NAS, advanced endoscopy training programs should utilize competency based medical education and demonstrate that advanced endoscopy trainees (AETs) have attained the technical and cognitive skills required for safe and effective unsupervised practice in advanced endoscopy. Based on the investigators research, the investigators can draw two conclusions: a) individuals in training in any technical procedure acquire skills at different rates and emphasis needs to be shifted away from the number of procedures performed to performance metrics with defined and validated competency thresholds of performance and b) current guidelines of performing 150 EUS and 180 ERCPs are inadequate to achieve competence in EUS and ERCP, respectively. With the expanding indications and applications of EUS and ERCP and establishment of a number of "third tier" training programs in advanced endoscopy, standardization of the performance of EUS and ERCP and definition of competence and training among AETs is of paramount importance. The potential impacts of this study's results are multifold: i) facilitate the ability of training programs to evolve with the new ACGME/NAS reporting requirements, (ii) help program directors/trainers and trainees identify specific skill deficiencies in training and allowing for tailored, individualized remediation, (iii) create a centralized national database that would allow generation of "on-demand" detailed reports on how individual trainees are progressing compared with their peers across the nation, (iv) establish reliable and generalizable standardized learning curves (milestones) and competency benchmarks that national GI societies and training programs can use to develop credentialing guidelines.

APPROACH AND RESEARCH STRATEGY Setting and Subject Recruitment: Program directors and AETs at all advanced endoscopy programs registered with the ASGE will be invited to participate in this study and will be considered as study participants. AETs will complete a questionnaire to determine baseline characteristics and prior experience with EUS and ERCP. AETs' prior experience with EUS and ERCP will not be an exclusion criterion for this study.

Competency assessment tools: Previous competency assessment tools have focused primarily on a limited number of motor skills involved in EUS and ERCP with no procedure-related cognitive skill assessment. The investigators have designed a prospective comprehensive competency assessment tool using validated benchmarks to define competency thresholds. The EUS and ERCP Skills Assessment Tool (TEESAT) can be used in a continuous fashion throughout the duration of training to grade technical and cognitive skills in EUS and ERCP in a balanced manner.

Learning curves during independent practice and Quality Indicators in EUS and ERCP: The ASGE and ACG Task Force on Quality in Endoscopy recently published documents highlighting quality indicators in EUS and ERCP. Impact of structured feedback on learning curves, specifically related to quality metrics, during the first year of independent practice for AETs has not been evaluated. This is an important component of construct validity for the proposed assessment tool and novel web-based comprehensive data collection and reporting, was identified as a priority research question by the Task Force. The defined performance targets and quality metrics will serve as benchmarks for analysis during training and first year of independent practice.

ELIGIBILITY:
Inclusion Criteria:

* Program directors and AETs at all advanced endoscopy programs registered with the ASGE will be invited to participate in this study and will be considered as study participants.

Exclusion Criteria:

* N/A

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Program directors and AETs at all advanced endoscopy programs registered with the ASGE will be invited to participate in this study and will be considered as study participants.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2015-07; Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Overall competency | Up to 12 months
  The proportion of advanced endoscopy trainees (AETs) that achieve overall competency in EUS and ERCP using a standardized competency assessment tool with a comprehensive data collection and reporting system.

SECONDARY OUTCOMES:
Number of advanced endoscopy fellows that reach competency | Up to 12 months
  Creation of a nationalized database utilizing the comprehensive assessment tool as to have advanced endoscopy fellows compare themselves to the national average in EUS and ERCP exams.

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Wani, MD, Principal Investigator — University of Colorado, Denver

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wani S, Han S, Simon V, Hall M, Early D, Aagaard E, Abidi WM, Banerjee S, Baron TH, Bartel M, Bowman E, Brauer BC, Buscaglia JM, Carlin L, Chak A, Chatrath H, Choudhary A, Confer B, Cote GA, Das KK, DiMaio CJ, Dries AM, Edmundowicz SA, El Chafic AH, El Hajj I, Ellert S, Ferreira J, Gamboa A, Gan IS, Gangarosa L, Gannavarapu B, Gordon SR, Guda NM, Hammad HT, Harris C, Jalaj S, Jowell P, Kenshil S, Klapman J, Kochman ML, Komanduri S, Lang G, Lee LS, Loren DE, Lukens FJ, Mullady D, Muthusamy RV, Nett AS, Olyaee MS, Pakseresht K, Perera P, Pfau P, Piraka C, Poneros JM, Rastogi A, Razzak A, Riff B, Saligram S, Scheiman JM, Schuster I, Shah RJ, Sharma R, Spaete JP, Singh A, Sohail M, Sreenarasimhaiah J, Stevens T, Tabibian JH, Tzimas D, Uppal DS, Urayama S, Vitterbo D, Wang AY, Wassef W, Yachimski P, Zepeda-Gomez S, Zuchelli T, Keswani RN. Setting minimum standards for training in EUS and ERCP: results from a prospective multicenter study evaluating learning curves and competence among advanced endoscopy trainees. Gastrointest Endosc. 2019 Jun;89(6):1160-1168.e9. doi: 10.1016/j.gie.2019.01.030. Epub 2019 Feb 7. PMID 30738985
- [Derived] Wani S, Keswani RN, Han S, Aagaard EM, Hall M, Simon V, Abidi WM, Banerjee S, Baron TH, Bartel M, Bowman E, Brauer BC, Buscaglia JM, Carlin L, Chak A, Chatrath H, Choudhary A, Confer B, Cote GA, Das KK, DiMaio CJ, Dries AM, Edmundowicz SA, El Chafic AH, El Hajj I, Ellert S, Ferreira J, Gamboa A, Gan IS, Gangarosa LM, Gannavarapu B, Gordon SR, Guda NM, Hammad HT, Harris C, Jalaj S, Jowell PS, Kenshil S, Klapman J, Kochman ML, Komanduri S, Lang G, Lee LS, Loren DE, Lukens FJ, Mullady D, Muthusamy VR, Nett AS, Olyaee MS, Pakseresht K, Perera P, Pfau P, Piraka C, Poneros JM, Rastogi A, Razzak A, Riff B, Saligram S, Scheiman JM, Schuster I, Shah RJ, Sharma R, Spaete JP, Singh A, Sohail M, Sreenarasimhaiah J, Stevens T, Tabibian JH, Tzimas D, Uppal DS, Urayama S, Vitterbo D, Wang AY, Wassef W, Yachimski P, Zepeda-Gomez S, Zuchelli T, Early D. Competence in Endoscopic Ultrasound and Endoscopic Retrograde Cholangiopancreatography, From Training Through Independent Practice. Gastroenterology. 2018 Nov;155(5):1483-1494.e7. doi: 10.1053/j.gastro.2018.07.024. Epub 2018 Jul 26. PMID 30056094
- [Derived] Wani S, Keswani R, Hall M, Han S, Ali MA, Brauer B, Carlin L, Chak A, Collins D, Cote GA, Diehl DL, DiMaio CJ, Dries A, El-Hajj I, Ellert S, Fairley K, Faulx A, Fujii-Lau L, Gaddam S, Gan SI, Gaspar JP, Gautamy C, Gordon S, Harris C, Hyder S, Jones R, Kim S, Komanduri S, Law R, Lee L, Mounzer R, Mullady D, Muthusamy VR, Olyaee M, Pfau P, Saligram S, Piraka C, Rastogi A, Rosenkranz L, Rzouq F, Saxena A, Shah RJ, Simon VC, Small A, Sreenarasimhaiah J, Walker A, Wang AY, Watson RR, Wilson RH, Yachimski P, Yang D, Edmundowicz S, Early DS. A Prospective Multicenter Study Evaluating Learning Curves and Competence in Endoscopic Ultrasound and Endoscopic Retrograde Cholangiopancreatography Among Advanced Endoscopy Trainees: The Rapid Assessment of Trainee Endoscopy Skills Study. Clin Gastroenterol Hepatol. 2017 Nov;15(11):1758-1767.e11. doi: 10.1016/j.cgh.2017.06.012. Epub 2017 Jun 16. PMID 28625816